CLINICAL TRIAL: NCT06748339
Title: Gut Microbiome Dyspiosis in Colorectal Cancer Egyptian Patients
Brief Title: Gut Microbiome and Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Heliopolis University (Other)
Responsible Party: Principal Investigator, Sara mostafa ElAdawy, lecturer, Heliopolis University
Other Study IDs: HU.REC.H10-2024
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: CRC; microbiome
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extracted from fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- contol group: 6 healthy participants
  Interventions: Other: no intervention
- CRC group: 12 newly diagnosed CRC patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Colorectal cancer (CRC) is reported to be the third leading cause of cancer deaths worldwide, and its prevalence is steadily rising in developing countries. It can be considered a marker of socioeconomic development and a marker of significant changes in food habits and lifestyle. In Egypt, CRC represents the seventh most common cancer. It is the third most reported cancer in males and the fifth most common cancer in females. microbiome dysbiosis may be involved in the pathogensis and thus pose a therapeutic target

DETAILED DESCRIPTION:
Many reports suggested the role of westernized dietary lifestyles, including high consumption of red meats, animal fats, and cholesterol-rich foods, as well as smoking, decreased physical activity, obesity, diabetes, alcohol consumption, or smoking, in CRC development. These changes in lifestyle are called the external factors, which are now linked to changes in the inner gut microenvironments, mainly the microbiomes. Our aim is to investigate the the changes in microbiome profile in relation to clinical, pathological and lifestyle factors

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 years to 80 years
* Patients with a newly diagnosed CRC

Exclusion Criteria:

* Patients with previously known CRC
* Pregnancy or Lactation
* Abdominal surgery within/up to 6 months prior to sample collection
* Antibiotics, corticosteroids, or probiotics up to three months prior to sample collection
* History of other types of cancer
* Subjects on a special diet
* Diabetes, liver, or kidney diseases
* CRC patients who used enema or underwent colonoscopy up to one week before sample collection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 newly diagnosed CRC patiens vs 6 healthy voulnteers
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
The effect of food and lifestyle on microbiome | "through study completion, an average of 1 year"
  correlation between food and lifestyle with microbiome profiles
microbiome profile and CRC pathogensis | "through study completion, an average of 1 year"
  correlation between microbiome profile and CRC pathogensis

CONTACTS AND LOCATIONS:
Overall Officials: sara M eladwy, Principal Investigator — Heliopolis University
Locations (1):
- cairo university Hopitals (elKasr ELieny ), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Patients' information will be assigned codes. no need to reveal it

REFERENCES:
- [Background] Baas FS, Brusselaers N, Nagtegaal ID, Engstrand L, Boleij A. Navigating beyond associations: Opportunities to establish causal relationships between the gut microbiome and colorectal carcinogenesis. Cell Host Microbe. 2024 Aug 14;32(8):1235-1247. doi: 10.1016/j.chom.2024.07.008. PMID 39146796
- See also: Navigating beyond associations: Opportunities to establish causal relationships between the gut microbiome and colorectal carcinogenesis — https://pubmed.ncbi.nlm.nih.gov/39146796/